CLINICAL TRIAL: NCT06272214
Title: The Role of Adjuvant Radiotherapy in the Treatment for Resectable Locally Advanced Esophageal Squamous Cell Carcinoma After Neoadjuvant Chemotherapy Combined With Immunotherapy: A Multi-center, Phase II Randomized Clinical Study
Brief Title: Adjuvant Radiotherapy for Esophageal Squamous Cell Carcinoma in the Era of Immunotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yang Yang, Doctor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2024-048
Record Dates: First submitted 2024-02-04; First posted 2024-02-22 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Adjuvant Radiotherapy
Keywords: Esophageal cancer; Surgery; Neoadjuvant; Chemotherapy; Immunotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy, Adjuvant; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant radiotherapy (Experimental): Following surgery, patients start adjuvant radiotherapy 4-6 weeks after the operation, with a radiation dose of 45Gy/25F/5W, completed no later than 8 weeks post-surgery. Two weeks after completing radiotherapy, patients continue with immunotherapy maintenance therapy for up to 1 year (17 cycles Q3W) or until tumor progression.
  Interventions: Radiation: Adjuvant radiotherapy
- Observation (Active Comparator): Patients receive surgery after neoadjuvant chemotherapy combined with immunotherapy for esophageal cancer, followed by active survillance and maintenance therapy with PD1/PDL1 inhibitors for up to 1 year (17 cycles Q3W) or until tumor progression.
  Interventions: Other: Observation

INTERVENTIONS:
Radiation: Adjuvant radiotherapy — The start time for radiotherapy is 4-6 weeks after surgery, typically not exceeding 8 weeks. Intensity-modulated radiation therapy (IMRT) will be used, with a total dose of 45Gy administered in 25 fractions, five times per week.
  The recommended target delineation for radiotherapy is based on the Chinese guidelines for radiation therapy of esophageal cancer, which mainly covers the high-risk lymph node area.
  Arms: Adjuvant radiotherapy
Other: Observation — Patients receive surgery after neoadjuvant chemotherapy combined with immunotherapy for esophageal cancer, followed by active survillance and maintenance therapy with PD1/PDL1 inhibitors for up to 1 year or until tumor progression.
  Arms: Observation

SUMMARY:
This study is a multicenter, prospective, randomized phase II trial aimed at exploring the value of adjuvant radiotherapy in patients at high risk of recurrence after neoadjuvant chemoradiotherapy for esophageal cancer. The study primarily includes patients with esophageal cancer who underwent neoadjuvant chemoradiotherapy and surgery and did not achieve complete pathological response (non-pCR) postoperatively and were defined as preoperative clinical stage at T3-4N+M0.

Eligible patients will be randomized in a 1:1 ratio into two groups: the observation group and the adjuvant radiotherapy group. The control group consists of patients who receive surgery after neoadjuvant chemotherapy combined with immunotherapy for esophageal cancer, followed by maintenance therapy with PD1/PDL1 inhibitors for up to 1 year or until tumor progression. The adjuvant radiotherapy group receives additional adjuvant radiotherapy on top of the control group's treatment. The specific treatment process involves receiving 2 cycles of neoadjuvant chemotherapy combined with immunotherapy (PD1/PDL1 inhibitors) before potentially curative esophageal cancer surgery. The chemotherapy regimen includes paclitaxel in combination with platinum agents, with a preference for albumin-bound paclitaxel (280mg/m2 on Day 1, or 100mg on Days 1, 8, and 15) in combination with carboplatin (AUC=5). Following surgery, patients start adjuvant radiotherapy 4-6 weeks after the operation, with a radiation dose of 45Gy/25F/5W, completed no later than 8 weeks post-surgery. Two weeks after completing radiotherapy, patients continue with immunotherapy maintenance therapy for up to 1 year or until tumor progression. Subsequently, follow-up visits are scheduled every 3-4 months for the first 3 years, every 6 months for the next 2 years, and annually thereafter. The primary endpoint is 2-year disease-free survival (DFS), and secondary endpoints include overall survival (OS), local recurrence-free survival (LRFS), distant metastasis-free survival (DMFS), recurrence patterns, and safety assessment. Additionally, the study will explore biomarkers predicting treatment efficacy and adverse reactions in subjects, including PD-L1 expression, ctDNA clearance status, infiltrating immune cell types and quantities, cytokine expression, and other tumor biomarkers. This exploration aims to guide stratified precision treatment for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and voluntarily sign the written informed consent form, which must be signed before the specified research procedures required by the study are performed.
2. Subjects in this study are male or female aged ≥18 and ≤75 years at the time of signing the informed consent form.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 or Karnofsky Performance Status (KPS) score ≥80 points (see Table 1) at the time of signing the informed consent form.
4. Histologically confirmed esophageal squamous cell carcinoma.
5. The initial patient is a resectable or potentially resectable cT3-4N0 or T1-4N+ patient (AJCC 8th edition) who underwent 2 cycles of neoadjuvant immunotherapy and chemotherapy followed by surgical R0 resection, with postoperative pathology not achieving complete response (non-pCR).
6. Good organ function as determined by the following requirements: a. Hematology (without blood component or growth factor support within 7 days prior to the start of study treatment): i. Absolute neutrophil count (ANC) ≥1.5×109/L (1500/mm3). ii. Platelet count ≥100×109/L (100,000/mm3). iii. Hemoglobin ≥90g/L. b. Renal: i. Calculated creatinine clearance rate (CrCl) ≥50 mL/min. * CrCl will be calculated using the Cockcroft-Gault formula: CrCL (mL/min) = {(140 - age) × weight (kg) × F} / (SCr (mg/dL) × 72) where F = 1 for males and F = 0.85 for females; SCr = serum creatinine. ii. Urinary protein < 2+ or 24-hour urinary protein quantitation < 1.0 g. c. Hepatic: i. Total bilirubin (TBiL) ≤1.5×ULN. ii. AST and ALT ≤2.5×ULN; for subjects with liver metastasis, AST and ALT can be ≤5×ULN. iii. Serum albumin (ALB) ≥28 g/L. d. Coagulation function: International Normalized Ratio (INR) and activated partial thromboplastin time (APTT) ≤1.5×ULN (unless the subject is receiving anticoagulant therapy, and INR and APTT are within the expected range for anticoagulant therapy). e. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%.
7. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 3 days before the first dose (if urine pregnancy test results cannot be confirmed as negative, a serum pregnancy test must be performed, and serum pregnancy test results will be used) and agree to use highly effective contraception continuously for 120 days after the last dose of study drug; the decision to stop contraception after this time point should be discussed with the investigator.
8. Male subjects who are not surgically sterile and who are sexually active with female partners of childbearing potential must use effective contraception continuously from the screening period through 120 days after the last dose; the decision to stop contraception after this time point should be discussed with the investigator.
9. Subjects are willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study requirements.

Exclusion Criteria:

1. Stage IV metastatic esophageal cancer patients with initial diagnosis of metastasis to visceral organs (such as liver, bone, lung, brain, adrenal gland, etc.).
2. Patients who did not achieve R0 resection after surgery, including R1 and R2 resection.
3. Patients who achieved complete pathological response (pCR) after surgery.
4. Patients with a history of chest radiation therapy.
5. Patients with esophagomediastinal fistula and/or esophagotracheal fistula before treatment.
6. Pregnant or lactating female patients.
7. Patients who cannot provide informed consent due to psychological, family, social, or other reasons.
8. Patients with a history of malignant tumors other than esophageal cancer before enrollment, unless it is non-melanoma skin cancer, in situ cervical cancer, or cured early-stage prostate cancer.
9. Patients who cannot tolerate chemotherapy or radiation therapy due to severe heart, lung, liver, kidney dysfunction, cachexia, etc.
10. Patients with active autoimmune diseases, a history of autoimmune diseases (including but not limited to colitis, hepatitis, hyperthyroidism, etc.), a history of immunodeficiency (including HIV-positive test results), or other acquired or congenital immunodeficiency diseases, organ transplantation, or allogeneic bone marrow transplantation history.
11. Patients with active hepatitis B (HBV DNA ≥ 2000 IU/mL or 10×4 copies/mL), hepatitis C (positive hepatitis C antibody, with hepatitis C virus RNA (HCV-RNA) level higher than the detection limit).
12. Patients with a history of immunodeficiency diseases; HIV antibody-positive individuals; those currently using systemic corticosteroids or other immunosuppressive agents for an extended period.
13. Severe infections occurring within 4 weeks before the first dose, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia; active infections treated with systemic anti-infective therapy within 2 weeks before the first dose (excluding antiviral therapy for hepatitis B or hepatitis C).
14. Known active tuberculosis (TB) or suspected active TB subjects, who should undergo clinical examination for exclusion; known active syphilis infection.
15. Vaccination with live vaccines or attenuated live vaccines within 30 days before the first dose, or planned vaccination with live vaccines or attenuated live vaccines during the study period, with the use of inactivated vaccines allowed.
16. A history of interstitial lung disease or non-infectious pneumonitis.
17. A history of myocarditis, cardiomyopathy, malignant arrhythmias. Patients with unstable angina, myocardial infarction, congestive heart failure (New York Heart Association Functional Classification ≥2) or vascular diseases (such as aortic aneurysms at risk of rupture) within 12 months before the first dose or other cardiac injuries that may affect the safety assessment of the study drug (such as poorly controlled arrhythmias, myocardial ischemia).
18. Known psychiatric illness, substance abuse, alcoholism, or drug abuse history.
19. Local or systemic diseases not caused by malignant tumors; or diseases or symptoms secondary to tumors, which may lead to a higher medical risk and/or uncertainty in survival assessment, such as tumor lysis reaction (white blood cell count > 20×109/L), cachexia presentation (weight loss > 10% in the 3 months before screening), etc.
20. Any condition considered by the investigator as posing a risk to the subject, interfering with the evaluation of the study drug, or affecting the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
2-year DFS | 24 months
  Time between enrollment and recurrence of disease or death

SECONDARY OUTCOMES:
OS | occurence or end of follow-up（2 years after enrollment）, which comes first
  Overall survival，Time between enrollment and death
LRFS | 24 months
  Time between enrollment and local recurrence
DMFS | 24 months
  distant metastasis free survival,Time between enrollment and distant metastasis
HRQoL | 3 months, 1year, 2 years after surgery
  The EORTC QLQ-C30 questionnaire will be used. Scale scores will be calculated following the scoring guidelines of the EORTC questionnaires. Scores will be summarized by means of the appropriate descriptive statistics (mean + SD or median + IQR) at each measurement point.
Adverse effects recorded during radiotherapy and PD1/PDL1 inhibitors maintaince period | occurence or end of follow-up（2 years after enrollment), which comes first
  safety
Incidence of Recurrence | occurence or end of follow-up（2 years after enrollment), which comes first
  including local recurrence and distant metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Youhua Jiang, M.D., Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Kelly RJ, Ajani JA, Kuzdzal J, Zander T, Van Cutsem E, Piessen G, Mendez G, Feliciano J, Motoyama S, Lievre A, Uronis H, Elimova E, Grootscholten C, Geboes K, Zafar S, Snow S, Ko AH, Feeney K, Schenker M, Kocon P, Zhang J, Zhu L, Lei M, Singh P, Kondo K, Cleary JM, Moehler M; CheckMate 577 Investigators. Adjuvant Nivolumab in Resected Esophageal or Gastroesophageal Junction Cancer. N Engl J Med. 2021 Apr 1;384(13):1191-1203. doi: 10.1056/NEJMoa2032125. Erratum In: N Engl J Med. 2023 Feb 16;388(7):672. doi: 10.1056/NEJMx220014. PMID 33789008
- [Background] Luo H, Lu J, Bai Y, Mao T, Wang J, Fan Q, Zhang Y, Zhao K, Chen Z, Gao S, Li J, Fu Z, Gu K, Liu Z, Wu L, Zhang X, Feng J, Niu Z, Ba Y, Zhang H, Liu Y, Zhang L, Min X, Huang J, Cheng Y, Wang D, Shen Y, Yang Q, Zou J, Xu RH; ESCORT-1st Investigators. Effect of Camrelizumab vs Placebo Added to Chemotherapy on Survival and Progression-Free Survival in Patients With Advanced or Metastatic Esophageal Squamous Cell Carcinoma: The ESCORT-1st Randomized Clinical Trial. JAMA. 2021 Sep 14;326(10):916-925. doi: 10.1001/jama.2021.12836. PMID 34519801
- [Background] van den Ende T, de Clercq NC, van Berge Henegouwen MI, Gisbertz SS, Geijsen ED, Verhoeven RHA, Meijer SL, Schokker S, Dings MPG, Bergman JJGHM, Haj Mohammad N, Ruurda JP, van Hillegersberg R, Mook S, Nieuwdorp M, de Gruijl TD, Soeratram TTD, Ylstra B, van Grieken NCT, Bijlsma MF, Hulshof MCCM, van Laarhoven HWM. Neoadjuvant Chemoradiotherapy Combined with Atezolizumab for Resectable Esophageal Adenocarcinoma: A Single-arm Phase II Feasibility Trial (PERFECT). Clin Cancer Res. 2021 Jun 15;27(12):3351-3359. doi: 10.1158/1078-0432.CCR-20-4443. Epub 2021 Jan 27. PMID 33504550
- [Background] Yin J, Yuan J, Li Y, Fang Y, Wang R, Jiao H, Tang H, Zhang S, Lin S, Su F, Gu J, Jiang T, Lin D, Huang Z, Du C, Wu K, Tan L, Zhou Q. Neoadjuvant adebrelimab in locally advanced resectable esophageal squamous cell carcinoma: a phase 1b trial. Nat Med. 2023 Aug;29(8):2068-2078. doi: 10.1038/s41591-023-02469-3. Epub 2023 Jul 24. PMID 37488287
- [Background] Matsuda S, Kawakubo H, Okamura A, Takahashi K, Toihata T, Takemura R, Mayanagi S, Hirata K, Irino T, Hamamoto Y, Takeuchi H, Facs, Watanabe M, Kitagawa Y. Distribution of Residual Disease and Recurrence Patterns in Pathological Responders After Neoadjuvant Chemotherapy for Esophageal Squamous Cell Carcinoma. Ann Surg. 2022 Aug 1;276(2):298-304. doi: 10.1097/SLA.0000000000004436. Epub 2020 Oct 16. PMID 33074909
- [Background] Yang Y, Liu J, Liu Z, Zhu L, Chen H, Yu B, Zhang R, Shao J, Zhang M, Li C, Li Z. Two-year outcomes of clinical N2-3 esophageal squamous cell carcinoma after neoadjuvant chemotherapy and immunotherapy from the phase 2 NICE study. J Thorac Cardiovasc Surg. 2024 Mar;167(3):838-847.e1. doi: 10.1016/j.jtcvs.2023.08.056. Epub 2023 Sep 9. PMID 37696429